CLINICAL TRIAL: NCT00246584
Title: Long-Term Treatment, Multicenter, Open-Label Study With SPP100 in Patients With Essential Hypertension
Brief Title: A Long Term Study of SPP100 in Patients With Essential Hypertension (Trial is Not Recruiting in the US)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPP100A1202
Record Dates: First submitted 2005-10-27; First posted 2005-10-31 (Estimated); Last update posted 2006-07-28 (Estimated); Status verified 2006-07

CONDITIONS: Hypertension
Keywords: Hypertension; angiotensin; renin; aliskiren
MeSH Terms: conditions — Hypertension | interventions — aliskiren

INTERVENTIONS:
Drug: SPP100

SUMMARY:
This study will evaluate the safety and efficacy of long term treatment of SPP100 in patients with essential hypertension. (Trial is not recruiting in the US)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as essential hypertension -

Exclusion Criteria:

* Patients with secondary hypertension or suspected of having secondary hypertension.
* Patients suspected of having malignant hypertension
* Patients with any serious diseases or symptoms

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-10

PRIMARY OUTCOMES:
Incidence of adverse events, vital signs, abnormal laboratory changes,etc.

SECONDARY OUTCOMES:
Change from baseline in diastolic blood pressure after 52 weeks
Change from baseline in systolic blood pressure after 52 weeks
Diastolic blood pressure < 90 mmHg or a reduction of > 10 mmHg after 52 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharmaceuticals, Basel, Switzerland